CLINICAL TRIAL: NCT01068184
Title: A Phase I, Randomised, Double-Blind, Placebo-Controlled, 3-Part Study to Assess the Safety, Tolerability and Pharmacokinetics of Single and Multiple Oral Doses of AZD6553 in Healthy Volunteers (Parts A and B) and Patients (Part C) With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of of AZD6553 in Healthy Volunteers and Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: temporary hold in May 2010 due to an emerging PK profile that could not be aligned to the known pharmaceutical properties of the IMP (AZD6553).
Sponsor: AstraZeneca (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D2580C00001; 2009-016931-36 (EudraCT Number)
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: AZD6553; Chronic; obstructive; pulmonary; lung; respiratory disease; placebo-controlled; COPD; Healthy Volunteers; COPD Patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiolitis Obliterans Syndrome; Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: AZD6553
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6553 — Single or multiple oral dose
  Arms: 1
Drug: Placebo — single or multiple oral dose
  Arms: 2

SUMMARY:
AZD6553 is a new drug being developed as a possible treatment for patients with chronic obstructive pulmonary disease (COPD). COPD refers to chronic bronchitis and emphysema, a pair of two commonly co-existing diseases of the lungs in which the airways become inflamed and the small airsacs of the lungs become damaged. This leads to a limitation of the flow of air to and from the lungs causing shortness of breath. In contrast to asthma, the limitation of airflow is poorly reversible and usually gets progressively worse over time. There is an urgent medical need for therapies that could slow disease progression by targeting the underlying mechanisms associated with the changes in the lungs in patients with COPD. AZD6553 acts by reducing the activity of a protease found to be involved in the disease process in COPD. AZD6553 is being developed as a novel oral treatment to control the symptoms and exacerbations of COPD, and reduce the progression and severity of the disease. The purpose of this research study is to determine how safe and well-tolerated AZD6553 is and how much AZD6553 enters blood circulation by collecting blood and urine samples during the study. We are also investigating what AZD6553 is broken down into, when given orally, how much of the drug is cleared from the body via the kidneys, and the effect of taking the drug after food. This will all be done by analysis of blood and urine samples taken at various point during the study.

ELIGIBILITY:
Inclusion Criteria:

* Parts A and B only; Body mass index (BMI) between 18 and 30 kg/m2.
* Parts A and B only; Normal physical examination, laboratory values, and vital signs (blood pressure and pulse) unless the investigator considers an abnormality to be clinically irrelevant.
* Part C only; clinical diagnosis of COPD for at least one year and Post-bronchodilator FEV1 30 - 80% predicted, FEV1/FVC ratio < 70%

Exclusion Criteria:

* Participation in any clinical study with an investigational drug or new formulation of a marketed drug in the 3 months prior to Visit 2, or participation in a method development study one month prior to Visit 1
* Part C only: An acute exacerbation or acute respiratory infection (upper or lower) in the 4 weeks prior to Visit 1 or Visit 2.
* Part C only: Concomitant diagnosis of significant pulmonary disease other than COPD, including symptomatic asthma, cystic fibrosis and allergic bronchopulmonary aspergillosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety variables (adverse events, ECG's blood pressure, pulse, safety lab) | Part A Intensive sampling for 24 hours , frequent sampling up to 72 hours, Part B Frequent Sampling over 12 days with intensive sampling on Days 1-2 and 8-9
Pharmacokinetic variables:-Cmax, AUC, tmax and t1/2 | Part A Intensive sampling for 24 hours , frequent sampling up to 72 hours, Part B Frequent Sampling over 12 days with intensive sampling on Days 1-2 and 8-9

SECONDARY OUTCOMES:
Lung Function SVC, IC, FEV1, FVC | Part C Days 2, 7 and 14
Pharmacokinetic variables; Urine CLR | Part A Days 1 and 2, Part B, Days 1 and 2 and Days 8,9 and 10, and Part C Day 1 and Day 14

CONTACTS AND LOCATIONS:
Overall Officials: T G K Mant, FRCP (UK) FFPM, Principal Investigator — Quintiles Drug Research Unit at Guy's Hospital; Joanna Marks-Konczalik, Study Director — AstraZeneca R&D Charnwood
Locations (1):
- Research Site, London, United Kingdom